CLINICAL TRIAL: NCT05512026
Title: A Prospective, Pre-Market, Multicenter, Non-significant Risk Study to Validate the Performance of the Poseidon System for Fluid Management During Water-aided Colonoscopy
Brief Title: Performance of the Poseidon System for Fluid Management During Water-aided Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: WAE Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-0100
Record Dates: First submitted 2022-08-18; First posted 2022-08-23 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Colonic Disease
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Intervention Model Description: Up to 30 subjects Fifteen subjects will be enrolled in this study and undergo water-aided colonoscopy with the Poseidon System. If the Primary Endpoint and Secondary Endpoint 1 are achieved in the first 15 subjects, the study will be complete.
  If the Primary Endpoint or Secondary Endpoint 1 are not achieved, changes to the device design will be made and this protocol will be conducted again in a second group of 15 subjects with updated device.
Masking Description: Patients will be de identified and assigned a designated number for inclusion in case report forms. Source documents will contain patient information and assigned study participant number.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Feasibility Assessment (Experimental): The Poseidon System is investigational and indicated to provide a pathway to control waste fluid during irrigation of the colon. All consented patients will receive the Device use during their colonoscopy procedure.
  Interventions: Device: Feasibility Assessment

INTERVENTIONS:
Device: Feasibility Assessment — To validate the performance of the Poseidon System™ for fluid management during water-aided endoscopic procedures in the colon.

SUMMARY:
To validate the performance of the Poseidon System™ for fluid management during water-aided endoscopic procedures in the colon.

DETAILED DESCRIPTION:
The Poseidon System is a fluid management system that is investigationally indicated to provide a pathway to control waste fluid during irrigation of the colon. The Poseidon device is a manually placed and controlled device that provides support and sealing on the perimeter of an endoscope while managing fluids naturally exiting the anus, during a colonoscopy procedure. The device consists of a introducer and hand piece that allows for passage of an endoscope with valves and a retention balloon that minimize fluid passage with a single-use waste bag for collecting fluid and debris. The Poseidon™ System is not yet FDA 510(k) cleared.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or greater.
2. Patients that have an indication to undergo water-aided colonoscopy.
3. Subjects with the ability to understand the requirements of the study, who have provided written informed consent, and who are willing and able to return for the required follow-up assessments.

Exclusion Criteria:

1. Subject unable or unwilling to provide informed consent.
2. Subjects with prolapsing hemorrhoids that require intervention or hemorrhoids that have been treated within last 3 months.
3. Prior TAMIS (Trans-anal minimally invasive surgery) or TEMS (Trans-anal micro endoscopic surgery).
4. Any condition that in the opinion of the Investigator would create an unsafe clinical situation that would not allow the patient to safely undergo an endoscopic procedure.
5. Pregnant or lactating women or women of childbearing potential who do not employ a reliable method of contraception as judged by the Investigator, and/or are not willing to use reliable contraception for the duration of study participation.
6. Patient is enrolled in another trial that could interfere with the endpoint analyses of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-12 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Human Factors as assessed using the frequency of failure | 1 day
  The design of the Poseidon System meets all acceptance criteria for design validation.
  User is able to operate device per the instructions for use. This criterion will be assessed in a pass/fail manner with an allowance of only 1 failure in the first 15 subjects and 1 failure in the second 15 subjects (if applicable).
Colonoscope Control as assessed using a 5-point Likert scale from 1 (Strongly Disagree) to 5 (Strongly Agree). | 1 day
  User shall not adversely influence typical actuation of a scope during colonoscopy procedure as assessed using a 5-point Likert scale.
Device Usability 1 as assessed using a 5-point Likert scale from 1 (Strongly Disagree) to 5 (Strongly Agree). | 1 day
  User assessment of functional acceptability of Poseidon device ratchet location as assessed using a 5-point Likert scale.
Device Usability 2 as assessed using a 5-point Likert scale from 1 (Strongly Disagree) to 5 (Strongly Agree). | 1 day
  User assessment of functional acceptability of Poseidon device intergluteal cleft fit as assessed using a 5-point Likert scale
Fluid retention as assessed using a 5-point Likert scale from 1 (Strongly Disagree) to 5 (Strongly Agree). | 1 day
  The Poseidon System shall minimize passage of fluids through and around the scope lumen when a scope is in the device, as assessed using a 5-point Likert scale.

SECONDARY OUTCOMES:
Number of Adverse Events | 2 weeks
  Safety defined as the occurrence of all adverse events measured from the Index Procedure through the 2 Week Post Procedure Follow-up Visit.
Time measured in minutes | 1 day
  Procedure time measured in minutes from the point of scope insertion to the point of scope removal (scope-in / scope-out).
Number of Device Deficiencies | 1 day
  Device deficiencies defined as an inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance including malfunctions, use errors, and inadequate labelling.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Nettt, MD, Principal Investigator — Sutter Health
Locations (1):
- Sutter Health - 1101 Van Ness Ave, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Not applicable to this trial. Trial and device validation will be used to commercially release product only.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT05512026/Prot_SAP_001.pdf